CLINICAL TRIAL: NCT02730013
Title: The MIND-FUN Research Study: Mind-motor Exercise to Improve Cognition and Functional Fitness
Brief Title: Mind-motor Exercise to Improve Cognition and Functional Fitness
Acronym: MIND-FUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Schlegel Villages: Retirement Homes and Long Term Care (Unknown); University of Waterloo Research Institute for Aging (Unknown)
Responsible Party: Sponsor
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10012765
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2017-09

CONDITIONS: Cognitive Decline
Keywords: Older adults; Square stepping exercise; Mind-motor exercise; Long-term care; Global cognitive functioning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Square Stepping Exercise (Experimental): Square-Stepping Exercise (SSE) Intervention Participants in this group will attend a square-stepping exercise intervention 60 minutes: 5 minute for attendance, 5-10 minute warm-up 40-45 minute SSE and 5-10 minute cool-down, on two days a week for a duration of 12 weeks.
  Interventions: Behavioral: Square Stepping Exercise
- Usual-care wait-list control (No Intervention): This group will receive standard care and be invited to partake in the intervention after all assessments have been completed.

INTERVENTIONS:
Behavioral: Square Stepping Exercise — Square Stepping Exercise involves mimicking a stepping pattern demonstrated by an instructor. The stepping patterns become progressively difficult and involve forward, backward, lateral and diagonal movements on a 250cm long mat with 25cm square grids.
  In a group setting, an instructor will demonstrate walking patterns on a gridded mat to the participants and the participants must memorize and repeat the patterns on their own. This program has over 200 patterns that increase in difficulty from beginner to advanced. Eighty percent of the group must successfully complete the patterns to move onto the next pattern. Social engagement is encouraged.
  Other Names: Mind-motor exercise
  Arms: Square Stepping Exercise

SUMMARY:
This is a 3 month cluster randomized controlled trial using a square-stepping exercise program (a.k.a. mind-motor exercise) in retirement and long-term care residences to improve global cognitive functioning in older adults with and without cognitive impairments. The investigators intend this project to be pragmatic and therefore will include residents with dementia and walking aids if the participants wish to participate. The primary outcome is global cognitive functioning, secondary outcomes include: single and dual task gait (only completed with those without dementia), oculomotor functioning, and functional fitness. The investigators hypothesize that there will be improvements in primary and secondary outcomes in the intervention group.

DETAILED DESCRIPTION:
Square Stepping Exercise (SSE) can be best described as a visuospatial working memory task, with a stepping response and thus may be considered as a cognitive-physical exercise or alternatively as a type of mind-motor exercise. The SSE program was developed specifically to improve balance and lower extremity functioning and thereby prevent disability and institutionalization in older adults with recent evidence also suggesting that it may positively impact cognitive functioning.

Through the investigators' collaboration with Dr. Mike Sharratt, President of the Schlegel-University of Waterloo Research Institute for Aging, Jaimie Killingbeck, Program for Active Living Coordinator for Schlegel Villages, and Susan Brown, Research Coordinator for the Schlegel-University of Waterloo Research Institute for Aging this study aims to: further assess the feasibility of square-stepping exercise amongst older adults with a variety of cognitive abilities, increase our collaborative efforts in the broader community and to engage older adults in physical activity to improve global cognitive functioning through a mind-motor exercise intervention.

This study will be a cluster randomized controlled trial, stratified by long-term care or full continuum care of the 4 Schlegel Villages involved, not blinded. The investigators will stratify so that 1 long-term care and 1 full continuum will be randomized to begin the square-stepping program immediately, and 1 long-term care and 1 full continuum care will be randomized to usual-care wait list control group, that will begin the program once 12-week measurements are complete. The facilities were stratified to help balance baseline cognition between the intervention and control groups. The 4 facilities are: Long-term Care - Glendale Crossings and St. Claire; Full continuum Care - Tansley Woods and Winston Park. The sites were pre-randomized to allow facilities time to prepare their programming schedules to include square-stepping exercise to their residents. Intervention sites include Glendale Crossings and Tansley Woods and wait-list control sites include St. Claire and Winston Park. Outcomes assessments will be completed by graduate students and research assistants on this project. The assessments will be completed at each of the Villages. The Schlegel Villages staff Kinesiologists/ Exercise Therapists will implement the square-stepping exercise program during the 12 week period. Study staff will train the Schlegel Villages staff on how to implement the program.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the 4 Schlegel Villages: Glendale Crossing, St. Clair, Tansley Woods, Winston Park
* Both males and females

Exclusion Criteria:

* Wheelchair bound residents
* Residents who are blind or deaf without aids
* Any residents who may not be able to participate due to health or behaviours in collaboration and discretion of the Schlegel Villages staff.
* Residents who have a diagnosis of dementia, have a score of greater than 3 on the Cognitive Performance Scale (determined by each Schlegel Village) and advice from Schlegel Villages staff will be excluded from specific assessments (dual-task gait; oculomotor function; global cognitive functioning outcomes; Montreal Cognitive Assessment; 2 cognitive questions).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Composite score from Cambridge Brain Sciences Cognitive Battery | Change from 0 to 12 weeks
  To assess global cognitive function.

SECONDARY OUTCOMES:
Gait variability (stride time) under dual-task conditions | Change from 0 to 12 weeks
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as the coefficient of variation of step length (SD/mean x100). Measured with GAITRite system.
Gait variability (stride time) under single-task conditions | Change from 0 to 12 weeks
  Gait variability is the stride-to-stride fluctuations of the way someone walks and will be calculated as the coefficient of variation of step length (SD/mean x100). Measured with GAITRite system (portable gait analysis).
Gait velocity (speed) under dual-task conditions | Change from 0 to 12 weeks
  Average walking speed (gait velocity) measured with the GAITRite system (portable gait analysis)
Gait velocity (speed) under single-task conditions | Change from 0 to 12 weeks
  Average walking speed (gait velocity) measured with the GAITRite system (portable gait analysis).
Step length (average) under dual-task conditions | Change from 0 to 12 weeks
  Mean step length calculated from GAITRite system (portable gait analysis).
Step length (average) under single-task conditions | Change from 0 to 12 weeks
  Mean step length calculated from GAITRite system (portable gait analysis).
Memory composite score | Change from 0 to 12 weeks
  Measured by Cambridge Brain Sciences - composite score from 4 memory tasks
Reasoning composite score | Change from 0 to 12 weeks
  Measured by Cambridge Brain Sciences - composite score from 3 reasoning tasks
Concentration composite score | Change from 0 to 12 weeks
  Measured by Cambridge Brain Sciences - composite score from 3 concentration tasks
Planning (executive functioning) composite score | Change from 0 to 12 weeks
  Measured by Cambridge Brain Sciences - composite score from 2 planning (executive function) tasks
Short Performance Physical Battery - Balance | Change from 0 to 12 weeks
  To assess balance measured by Side by Side Stand, Semi-Tandem Stand, Tandem Stand to obtain a balance test score.
Neuropsychiatric Inventory Questionnaire | change from 0 to 12 weeks
  To assess behavioural changes in residents with dementia

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petrella, MD, PhD, Principal Investigator — Western University
Locations (1):
- Western Centre for Public Health and Family Medicine, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No